CLINICAL TRIAL: NCT03369860
Title: Basi Neuro-cognitive Dell'Interazione Motoria
Brief Title: Neuro-cognitive Bases of Joint Action
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: JOINT
Record Dates: First submitted 2017-11-21; First posted 2017-12-12 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Health Behavior; Social Interaction
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Subjects (Experimental): Healthy Subjects take part in the experimental manipulation
  Interventions: Behavioral: Interactivity of Experimental Condition

INTERVENTIONS:
Behavioral: Interactivity of Experimental Condition — The neurofunctional correlates of motor control will be compared between a collaborative and non-interactive condition.

SUMMARY:
The ability to interact with conspecifics is crucial in life, yet there is no consensus on the underlying cognitive and neural mechanisms beyond those associated with imitative behaviors. This project aims to define a coherent model of non-imitative (complementary) motor interactions. The investigators hypothesize that these might be substantially based on the ability to integrate one's own and a partner's action within a unitary, dual- person (dyadic), motor plan that incorporates a shared goal.

With a novel "minimally-joint" paradigm the investigators will test this hypothesis and measure with behavioral measures (i.e., reaction times) whether the supposedly automatic tendency to imitate others is modulated by the need to coordinate with a partner to achieve a shared goal.

This paradigm will be also applied during a functional MRI experiment to describe the underlying neurophysiological patterns; using dynamic causal modeling the investigators will measure how the brain regions relevant for dyadic motor control are functionally linked.

This converging experimental strategy will permit to compare competing psychological and neural models of motor interactions in healthy participants, opening new experimental avenues for studies in adult neuropsychological patients and in children with typical and atypical social development.

ELIGIBILITY:
Inclusion Criteria:

* right handed; no contraindication to MRI

Exclusion Criteria:

* contraindication to MRI

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-12-20 (Estimated); Study Completion 2019-12-20 (Estimated)

PRIMARY OUTCOMES:
Reaction Times | 1 year
  The investigators will compare Reaction Times of participants recorded during Joint Action with those recorded in Non-Joint individual condition.
BOLD activations | 1 year
  The investigators will study the neurofunctional activations indexed by the Blood Oxygen Level Dependent (BOLD) recorded during Joint Action will be compared to the Non-Joint actions

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Galeazzi Orthopedic Hospital, Milan, Italy